CLINICAL TRIAL: NCT00779181
Title: A Phase 2, Dose-Ranging Study of the Safety and Efficacy of ADX415 Immediate-Release in the Treatment of Essential Hypertension
Brief Title: A Dose-Ranging Study of the Safety and Efficacy of ADX415 in the Treatment of Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Addrenex Pharmaceuticals, Inc. (Industry)
Responsible Party: Moise Khayrallah, PhD / President and CEO, Addrenex Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX415-301
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension
Keywords: Hypertension; High blood pressure; Htn; Addrenex
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ADX415 (high dose) (Experimental): A high dose of ADX415
  Interventions: Drug: ADX415
- ADX415 (mid level dose) (Experimental): A mid level dose of ADX415
  Interventions: Drug: ADX415
- ADX415 (low dose) (Experimental): A low dose of ADX415
  Interventions: Drug: ADX415
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX415 — ADX415 taken three times a day to achieve a high total daily dose
  Arms: ADX415 (high dose)
Drug: ADX415 — ADX415 taken three times a day to achieve a mid level total daily dose
  Arms: ADX415 (mid level dose)
Drug: ADX415 — ADX415 taken three times a day to achieve a low total daily dose
  Arms: ADX415 (low dose)
Drug: Placebo — Placebo taken three times a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine a safe and effective dose of ADX415 for the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hypertension
* Age 18-75 years, inclusive

Exclusion Criteria:

* Clinically significant illnesses or abnormalities upon evaluation
* Current treatment with 3 or more antihypertensive meds
* Presence of Type I or uncontrolled Type II diabetes
* Presence of alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in ABPM measures | Baseline to Day 26

SECONDARY OUTCOMES:
Treatment emergent adverse events, lab tests, vitals signs, and ECGs | Throughout treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Moise Khayrallah, PhD, Study Director — Addrenex Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Austin, Texas
  - San Antonio, Texas